CLINICAL TRIAL: NCT02585999
Title: The Pharmacokinetics of 12 Week Continuous Patch Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Antonella Lavelanet, Physician, Boston Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-34252
Record Dates: First submitted 2015-10-20; First posted 2015-10-26 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Pharmacokinetics
Keywords: Hormonal contraception, hormone pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Xulane (Other): All participants using the Xulane contraceptive patch for 12 continuous weeks
  Interventions: Device: Xulane Contraceptive Patch

INTERVENTIONS:
Device: Xulane Contraceptive Patch — Extended use (12 weeks) of contraceptive patch
  Other Names: Ortho Evra®

SUMMARY:
Investigators propose a descriptive pharmacokinetic study of the serum hormone levels of estrogen and progesterone with extended use (12 weeks) of the contraceptive patch. The primary objective is to assess the change in serum ethinyl estradiol (EE2) levels over 12 weeks of continuous contraceptive patch use. The secondary objective is assessing the the norelgestromin (NGMN) levels over the 12 weeks of continuous contraceptive patch use.

DETAILED DESCRIPTION:
For women who are seeking alternatives to long-acting contraceptives, the oral contraceptive pill and the contraceptive ring are often prescribed in an extended manner (12 weeks straight). The contraceptive patch, however, is not routinely prescribed in this way. Concerns have been raised that hormone levels, in particular estrogen, are higher among patch users than those who use oral contraception or the vaginal ring and that this may contribute to an increased risk of clot. However, few studies have actually looked at these hormone levels in women with extended use of the contraceptive patch.

The investigators plan to enroll eligible women age 18-39 who are willing to use the contraceptive patch continuously for twelve weeks, and can adhere to the study requirements for follow-up. All participants will have weekly serum assessments of ethinyl estradiol and norelgestromin levels. The investigators will enroll 30 women, in anticipation of a 33% attrition rate, with the goal of obtaining completed data on 20 participants. The study duration for an individual participant will be 12 weeks and the duration of the entire study will be one year.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to come to the clinic to have blood drawn weekly for 12 weeks, biweekly during weeks 4, 8, and 12, and for 3 days after the final patch is removed for blood draws for a total of 18 blood draws
* Willing and able to abstain from using any other hormonal contraceptive method while in the study and for the week prior to starting the study

Exclusion Criteria:

* Body Mass Index greater than 35
* Personal or Family History of Venothromboembolism
* Personal History of Migraines with Aura
* Personal History of Migraines without Aura
* Tobacco use greater than or equal to 15 cigarettes per day
* Current Pregnancy
* History of or Current Diagnosis of Cancer

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Lavelanet, DO, JD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 30 participants completed the baseline questionnaire, but 2 withdrew prior to starting the study.
Groups:
- Xulane: Participants exposed to contraceptive patch, Xulane.
  Xulane Contraceptive Patch (generic version of Ortho Evra®*): Extended use (12 Weeks) of Contraceptive Patch
Period: Overall Study
Arm/Group | Xulane
Started | 28
Completed | 26 (28 participants enrolled; 2 withdrew prior to starting, leaving 26 to complete study activity.)
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: 30 participants completed the baseline questionnaire, but 2 withdrew prior to starting the study.
Arm/Group | Xulane
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 13
  More than one race | 5
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum EE2 Levels Over 12 Weeks of Continuous Contraceptive Patch Use
Description: Liquid chromatography-tandem triple quadrupole mass spectrometry was utilized to assess EE2
Time Frame: Total of 18 blood draws - once at the end of each patch week and two times during weeks four, eight and twelve (with the additional blood draw occurring mid-week); and blood draws performed for three continuous days after the final patch was removed
Population: Analysis was performed on all samples. Thus samples for 28 participants were analyzed, including the one participant who began the study but withdrew early [lost to follow up]. The first blood draw occurred at the end of the first patch week; there was no baseline draw prior to patch use.
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Xulane: Participants exposed to Xulane Contraceptive Patch for 12 weeks of continuous use
Arm/Group | Xulane
Number analyzed (Participants) | 28
pg/ml
  Week 1 (end) | 12.5 (14.2)
  Week 2 (end) | 14.3 (23.9)
  Week 3 (end) | 10.9 (13.6)
  Week 3.5 (mid-week) | 42.9 (46.8)
  Week 4 (end) | 25.9 (33.7)
  Week 5 (end) | 34.1 (25.7)
  Week 6 (end) | 36.7 (34.1)
  Week 7 (end) | 24.7 (26.5)
  Week 7.5 (mid-week) | 48 (47.6)
  Week 8 (end) | 32.8 (30.7)
  Week 9 (end) | 40.7 (33.7)
  Week 10 (end) | 42.6 (31.4)
  Week 11 (end) | 41.2 (34)
  Week 11.5 (mid-week) | 47.1 (35.3)
  Week 12 (end) | 27 (27.7)
  Week 12.1 (day 1 post patch) | 17.8 (28.7)
  Week 12.2 (day 2 post patch) | 12 (17.4)
  Week 12.3 (day 3 post patch) | 10.4 (16.6)

2. Secondary Outcome: NGMN Levels Over 12 Weeks of Continuous Patch Use
Description: Liquid chromatography-tandem triple quadrupole mass spectrometry was utilized to assess NGMN
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Xulane
Number analyzed (Participants) | 28
ng/ml
  Week 1 (end) | 0.691 (0.279)
  Week 2 (end) | 0.699 (0.366)
  Week 3 (end) | 0.674 (0.275)
  Week 3.5 (mid-week) | 1.09 (0.436)
  Week 4 (end) | 0.746 (0.364)
  Week 5 (end) | 0.877 (0.549)
  Week 6 (end) | 0.913 (0.463)
  Week 7 (end) | 0.689 (0.340)
  Week 7.5 (mid-week) | 1.06 (0.653)
  Week 8 (end) | 0.789 (0.517)
  Week 9 (end) | 0.814 (0.555)
  Week 10 (end) | 0.837 (0.548)
  Week 11 (end) | 0.792 (0.551)
  Week 11.5 (mid-week) | 0.954 (0.707)
  Week 12 (end) | 0.593 (0.491)
  Week 12.1 (day 1 post patch) | 0.422 (0.513)
  Week 12.2 (day 2 post patch) | 0.221 (0.292)
  Week 12.3 (day 3 post patch) | 0.163 (0.288)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the entire course of the study (October 2015 through June 2016).
Description: The at risk numbers represent the 28 participants who were enrolled in the study.
Arm/Group | Xulane
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Xulane (N=28)
Any Adverse Event (General disorders) | 0

LIMITATIONS AND CAVEATS:
It is difficult to compare our findings with those of previous studies, as previous studies have used other instrumentation and techniques in analysis of EE2. Serum analysis was also performed after all samples were collected from participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No